CLINICAL TRIAL: NCT03793465
Title: Pilot-Tart Cherry, Mitral Transcriptome and POAF Incidence
Brief Title: Pilot-Tart Cherry, Mitral Transcriptome, and POAF Incidence
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Cherry Marketing Institute, Dewitt MI (USA) (Unknown)
Responsible Party: Principal Investigator, Steven Bolling, Professor of Surgery, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HUM00145800
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Post-operative Atrial Fibrillation (POAF)

STUDY DESIGN:
Intervention Model Description: Single arm, open-label design. Commercial Montmorency tart cherry juice concentrate. Consumption - 2 servings (1 ounce or 2 tablespoon/serving) per day for three days before cardiac surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tart Cherry Concentrate (Experimental): Single arm, open-label design. Commercial Montmorency tart cherry juice concentrate. Servings (1 ounce or 2 tablespoon/serving) per day for three days
  Interventions: Dietary Supplement: tart cherry concentrate

INTERVENTIONS:
Dietary Supplement: tart cherry concentrate — Consume 2 servings (1 ounce or 2 tablespoon/serving) per day for three days before cardiac surgery

SUMMARY:
Assess impact of Tart Cherry Concentrate in cardiac surgical patients on POAF and related clinical and economic outcomes. Measure inflammation gene transcripts in cardiac tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Males and female patients (age 50-79) at the Mitral Valve Clinic/CVC undergoing elective cardiac surgery for mitral valve repair without the Cox MAZE procedure (MVR patients also undergoing CABG and/or tricuspid valve repair are also eligible)
2. In sinus rhythm (no pre-operative atrial fibrillation, no hx of AF)

Exclusion Criteria:

1. Age ≥ 80 years
2. Diagnosed pre-operative chronic or paroxysmal AF
3. Prior ablation procedure for AF
4. Previous cardiac surgery
5. Implanted pacemaker
6. Active smoker
7. Comorbidities such as congenital or cardiac re-operation
8. Use of antiarrhythmic agents
9. Active inflammatory or infectious disease or malignancy
10. Diagnosed autoimmune disease
11. Corticosteroid or other immunomodulatory or immunosuppressive medication
12. Known sensitivity to sorbitol
13. Known gastric sensitivity to acidic juices like orange juice

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-08 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Patient-reported tolerability score | One week
  Patients will complete a brief questionnaire regarding gastrointestinal status, using the Bristol Stool Form Scale
Efficacy as measured by total number of days in hospital within 60 days of surgery | 60 days
  Total number of days in hospital within 60 days of the index surgery
Efficacy as measured by altered (+/- 0.5 fold change) atrial transcript expression (mRNA) related to NFκB activation | 30 days
  Altered (+/- 0.5 fold change) atrial transcript expression (mRNA) related to NFκB activation

SECONDARY OUTCOMES:
Time to conversion to normal sinus rhythm | 30 days
  Perioperative time to conversion to normal sinus rhythm
Heart rhythm at hospital discharge | 30 days
  Heart rhythm at hospital discharge
Heart rhythm at 30 days | 30 days
  Heart rhythm at 30 days
Need for permanent pacemaker within 30 days of surgery | 30 days
  Need for permanent pacemaker within 30 days of surgery
Cerebrovascular thromboembolism [stroke, TIA] | 30 days
  Incidences (yes/no, total number) of Cerebrovascular thromboembolism [stroke, TIA]
Non-cerebrovascular thromboembolism | 30 days
  Incidences (yes/no, total number) of Non-cerebrovascular thromboembolism
Bleeding | 30 days
  Incidences (yes/no, total number) of Bleeding
Cerebrovascular events | 30 days
  Incidences (yes/no, total number) of Cerebrovascular events
Incidences of postoperative clinical events | 30 days
  Incidences (yes/no, total number) of Non-cerebrovascular events
Length of Hospital Stay | 60 days
  LOS [Index hospitalization]
Number of Re-hospitalization and ED visits | 60 days
  Number of Re-hospitalization and ED visits
Number of Outpatient Interventions | 60 days
  Number of Outpatient interventions
Total Costs for Hospital stay | 60 days
  Costs [incident hospital stay]

CONTACTS AND LOCATIONS:
Overall Officials: Steven F Bolling, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No